CLINICAL TRIAL: NCT06341101
Title: Timely Recovery After Subclinical Heart Failure (TREASURE Trial)
Brief Title: Timely Recovery After Subclinical Heart Failure
Acronym: TREASURE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Academisch Ziekenhuis Maastricht (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Zenab Mohseni, PI, Academisch Ziekenhuis Maastricht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-503135-33-00; 2022-503135-33-00 (Other: EU trial number)
Record Dates: First submitted 2024-02-26; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Heart Failure; Diastolic Dysfunction
Keywords: Pre-Eclampsia; hypertension; heart failure; treatment
MeSH Terms: conditions — Heart Failure; Pre-Eclampsia; Hypertension | interventions — Perindopril; Valsartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Perindopril 2 mg) (Experimental): Eligible subjects will be counselled and upon informed consent randomized for either medication or care as usual (i.e. no medication). After a complete cardiovascular assessment, medication will be initiated open-labeled (Perindopril 2 mg or no medication). In case of side effects Perindopril will be replaced by Valsartan 40 mg twice daily. A blood pressure below 120/80 mmHg is targeted. Blood pressure will be measured once per two weeks until the targeted blood pressure is achieved or until medication dosage has increased 4 times, corresponding Perindopril 10mg as maximum dosage or corresponding Valsartan 320mg (160 mg twice daily) as maximum dosage.
  Interventions: Drug: Perindopril
- Standard care group (i.e. no medication) (No Intervention): Eligible subjects will be counselled and upon informed consent randomized for either medication or care as usual (i.e. no medication).

INTERVENTIONS:
Drug: Perindopril — In case of side effects Perindopril will be replaced by Valsartan
  Other Names: Valsartan
  Arms: Intervention group (Perindopril 2 mg)

SUMMARY:
The goal of this randomized controlled trial is to assess the effectiveness of ACE inhibitors versus standard care) in reversing asymptomatic heart failure (HF stage-B) and/or diastolic dysfunction during a two-year open-label treatment period for formerly preeclamptic women on:

1. Reversibility of structural and functional myocardial impairment in asymptomatic HF towards healthy values;
2. The progression from asymptomatic to symptomatic HF (symptoms scored based on the NYHA criteria);
3. Cardiovascular performance (volume- and pressure load), cardio metabolic risk factors (glucose metabolism, lipid status, kidney function) and quality of life (questionnaires);
4. Novel biomarkers and relevant microRNA's indicative for hypertrophy, fibrosis inflammation and ischemia.

Eligible subjects will be counselled and upon informed consent randomized for either medication group (n=65) or care as usual group (n=65). After a complete cardiovascular assessment, medication will be initiated open-labeled (Perindopril 2 mg or no medication). Thereafter, standard medical check-ups (blood pressure, ECG, kidney function, transthoracic cardiac ultrasound, endothelial function, quality of life questionnaires, medical history taking, blood and urine banking) will be performed every six months for two years.

Researchers will compare ACE inhibitor (Perindopril 2 mg) and care as usual (i.e. no medication) to investigate whether ACE inhibitor allows timely recovery after subclinical heart failure.

ELIGIBILITY:
Inclusion Criteria:

* All women who visit Maastricht Univeristy Medical Center+ for Cardiovascular screening with subclinical/asymptomatic heart failure (HF stage-B) and/or diastolic dysfunction;
* Aged 18 years and older;
* Premenopausal women with a history of preeclamptic pregnancy and premenopausal women with a history of normal pregnancy;
* Between 0.5 and 30 years postpartum;

Exclusion Criteria:

* Intention to pursue pregnancy within 2 years;
* Already using antihypertensive medication;
* Suffering diabetes mellitus, kidney failure (GFR<60 ml/min/1.73m2), pre-existent auto-immune disease and/or liver insufficiency;
* Breastfeeding during participation;
* Previous angio-edema

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-03-26 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
No left Ventricular Hypertrophy | From enrollment to the end of treatment after 2 years
  Left ventricular mass index <95 g/m2
No concentric remodeling | From enrollment to the end of treatment after 2 years
  Relative Wall Thickness ≤0.43
No impaired systolic function | From enrollment to the end of treatment after 2 years
  Left ventricular ejection fraction ≥55%
Normal diastolic function | From enrollment to the end of treatment after 2 years
  Septal e'≥8 and Lateral e'≥10 and Average e'≥9 and LA <34 cc/m2

CONTACTS AND LOCATIONS:
Locations (1):
- AZMaastricht, Maastricht, Limburg, Netherlands